CLINICAL TRIAL: NCT04650399
Title: A Multicenter, Randomized, Controlled, Double Blinded Pivotal Study to Evaluate Safety and Immunogenicity of a Live-attenuated Chikungunya Virus Vaccine Candidate (VLA1553) in Adolescents Aged 12 Years to <18 Years
Brief Title: A Multicenter Study to Evaluate Safety and Immunogenicity of a Live-attenuated Chikungunya Vaccine in Adolescents
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Butantan Institute (Other Government)
Collaborators: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VLA1553-321
Record Dates: First submitted 2020-11-25; First posted 2020-12-02 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-05

CONDITIONS: Chikungunya
MeSH Terms: conditions — Chikungunya Fever | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): VLA1553
  Interventions: Biological: Active
- Placebo (Placebo Comparator): Placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Active — Single intramuscular vaccination on Day 1 with VLA1553, a lyophilized live-attenuated Chikungunya vaccine candidate 1x10E4 TCID50 per dose
  Arms: Active
Biological: Placebo — Single intramuscular vaccination on Day 1 with Phosphate-Buffered Saline (PBS) as placebo
  Arms: Placebo

SUMMARY:
This is a prospective, randomized, double-blinded, multicenter, pivotal study evaluating the final dose of VLA1553 (1 x10E4 TCID50 per dose) in comparison to a placebo control. The final dose of VLA1553 or control will be administered as single immunization on Day 1. Overall, approximately 750 male and female subjects aged 12 years to <18 years will be enrolled into the study.

DETAILED DESCRIPTION:
This is a prospective, double-blinded, multicenter, randomized, pivotal Phase 3 study comprising approximately 750 subjects aged 12 years to <18 years randomized in a 2:1 ratio to the live-attenuated CHIKV vaccine candidate (VLA1553) or placebo. The final dose of lyophilized VLA1553 or placebo will be administered as a single intramuscular immunization. Subjects in this study will be stratified by baseline serostatus. The primary objective of the study is to evaluate the immunogenicity and safety of the adult dose of VLA1553 28 days following the single immunization. Immunogenicity evaluations in the immunogenicity subset will include the proportion of subjects with seroprotective neutralizing CHIKV antibody titers above a surrogate threshold indicative of protection. The surrogate of protection reasonably likely to predict clinical benefit has been established in non-human primate passive transfer studies using human sera from the Phase 1 study. Safety data collection and immunogenicity will continue to be assessed until Month 12.

ELIGIBILITY:
Inclusion Criteria:

1. From the 12th birthday to the last day before the 18th birthday on the Day of screening;
2. able to provide informed consent as well as written informed consent by the subject's legal representative ;
3. generally healthy as determined by the Investigator's clinical judgement based on medical history, physical examination and screening laboratory tests;
4. seropositive for previous CHIKV exposure (i.e. IgM+/IgG+ or IgM-/IgG+) or seronegative (i.e. IgM-/IgG-) as screened by CHIKV-specific ELISA.
5. for women of childbearing potential:

   1. negative serum or urine pregnancy test at screening.
   2. practiced an adequate method of contraception during 30 days before screening
   3. agrees to employ adequate birth control measures for the first three months post-vaccination (i.e. until Day 85).

Exclusion Criteria:

1. CHIKV infection in the past, including suspected CHIKV infection; is taking medication or other treatment for unresolved symptoms attributed to a previous CHIKV infection; or has participated in a clinical study involving an investigational CHIKV vaccine;
2. acute or recent infection;
3. tests positive for human immunodeficiency virus (HIV) human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV);
4. live virus vaccine within 28 days or inactivated vaccine within 14 days prior to vaccination in this study or plans to receive a vaccine within 28 days or 14 days after vaccination, respectively;
5. abnormal findings in any required study investigations (including medical history, physical examination, and clinical laboratory) considered clinically relevant by the Investigator which pose a risk for participation in the study;
6. medical history of or currently has acute or progressive, unstable or uncontrolled clinical conditions that pose a risk for participation in the study;
7. history of immune-mediated or clinically relevant arthritis / arthralgia;
8. history of malignancy in the past 5 years other than squamous cell or basal cell skin cancer. If there has been surgical excision or treatment more than 5 years ago that is considered to have achieved a cure, the subject may be enrolled;
9. known or suspected defect of the immune system, such as subjects with congenital or acquired immunodeficiency, including infection with HIV, status post organ transplantation or immuno-suppressive therapy within 4 weeks prior to vaccination;
10. history of any vaccine related contraindicating event (e.g., anaphylaxis, allergy to components of the candidate vaccine, other known contraindications);
11. with clinical conditions representing a contraindication to intramuscular vaccination and blood draws;
12. pregnant or lactating at the time of enrollment;
13. donation of blood, blood fractions or plasma within 30 days or received blood-derived products (e.g. plasma) within 90 days prior to vaccination in this study or plans to donate blood or use blood products until Day 180 of the study;
14. rash, dermatological condition or tattoos that would, in the opinion of the Investigator, interfere with injection site reaction rating;
15. known or suspected problem with alcohol or drug abuse as determined by the Investigator;
16. any condition that, in the opinion of the Investigator, may compromise the subjects well-being, might interfere with evaluation of study endpoints, or would limit the subject's ability to complete the study;
17. committed to an institution (by virtue of an order issued either by the judicial or the administrative authorities);
18. participation in another clinical study involving an investigational medicinal product (IMP) or device within 30 days prior to study enrollment or is scheduled to participate in another clinical study involving an IMP, or device during the course of this study;
19. member of the team conducting the study or in a dependent relationship with one of the study team members. Dependent relationships include close relatives (i.e., children, partner/spouse, siblings, parents) as well as employees of the Investigator or site personnel conducting the study.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 750 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2024-02-15 (Actual)

PRIMARY OUTCOMES:
Seroprotection | up to Day 29 after single vaccination
  Proportion of subjects with a seroprotective CHIKV antibody level determined by µPRNT (Micro Plaque Reduction Neutralization Test) for baseline negative subjects 28 days post-vaccination.

SECONDARY OUTCOMES:
Immunogenicity | until Day 8, Day 85, Day 180, and Month 12 after vaccination
  Immune response as measured by CHIKV-specific neutralizing antibody titers determined by μPRNT assay
Seroprotection up to 1 year | until Day 8, Day 29, Day 85, Day 180, and Month 12 after vaccination
  Proportion of subjects with seroprotective CHIKV antibody levels as determined by µPRNT Month 12.
Seroconversion up to 1 year | 12 months after vaccination
  Proportion of subjects with seroconversion as compared to baseline at Day 29, Month 6 and Month 12 as determined by μPRNT assay
Fold Increase in neutralizing antibodies | 12 months after vaccination
  Fold increase of CHIKV-specific neutralizing antibody titers determined by μPRNT assay at Days 8, 29, 85, 180 and at Month 12 post-vaccination as compared to baseline
Proportion of increase of neutralizing antibodies | 12 months after vaccination
  Proportion of subjects reaching an at least 4-fold, 8-fold, 16-fold or 64-fold increase in CHIKV-specific neutralizing antibody titer compared to baseline as measured by μPRNT assay
Immunogenicity per baseline serostatus | 12 months after vaccination
  Antibody titers, seroprotection and fold increases for CHIKV-specific neutralizing antibodies, determined by μPRNT assay at Days 1, 8, 29, 85, 180, and Month 12 post-vaccination stratified by baseline serostatus
Unsolicited adverse events | 6 months after vaccination
  Frequency and severity of unsolicited AEs until Day 29 and Month 6 post-vaccination
Solicited adverse reactions | 10 days after vaccination
  Frequency and severity of solicited injection site and systemic reactions within ten days post-vaccination
Frequency of adverse event of special interest | until 12 month after vaccination
  Frequency and severity of any Adverse Event of Special Interest
Viremia of vaccine strain | 29 days after vaccination
  Frequency of viremia of vaccine strain detected on Days 1 and 8 (and Day 29, if applicable) after vaccination
Frequency of Serious Adverse Event | until 12 month after vaccination
  Frequency and relatedness of any Serious Adverse Event (SAE) during the entire study period

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Boulos, MD, MSc, Study Chair — Butantan Institute; Valneva Austria GmbH, Study Director — Valneva Austria GmbH
Locations (10):
- Brazil (10):
  - CECOR - Centro Oncológico de Roraima, Boa Vista, Acre
  - Fundação de Medicina Tropical Dr. Heitor Vieira Dourado, Manaus, Amazonas
  - Núcleo de Medicina Tropical - Universidade Federal do Ceará, Fortaleza, Ceará
  - Associação Obras Sociais Irmã Dulce / Centro de Pesquisa Clínica - CPEC, Salvador, Estado de Bahia
  - Centro de Pesquisa e Desenvolvimento de Fármacos (CPDF) - Universidade Federal de Minas Gerais, Instituto de Ciências Biológicas, Belo Horizonte, Minas Gerais
  - Real Hospital Português de Beneficência em Pernambuco, Recife, Pernambuco
  - Centro de Pesquisas Clínicas Universidade Federal Sergipe, Aracaju, Sergipe
  - Faculdade de Medicina de São José do Rio Preto - FAMERP, São José do Rio Preto, São Paulo
  - Centro de Pesquisa Clínica da Faculdade de Medicina da Universidade Federal de Mato Grosso do Sul - UFMS, Campo Grande
  - Centro de Estudos do Instituto de Infectologia Emílio Ribas, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Buerger V, Pfeiffer A, Schoengrundner P, Seebacher J, Hochreiter R, Kosulin K, Zoihsl O, Weisova P, Mader R, Loch AP, Morandi E Jr, Nogueira ML, de Brito CAA, Croda J, Teixeira MM, Coelho IC, Gurgel R, da Fonseca AJ, de Lacerda MVG, Moreira ED Jr, Veiga APR, Eder-Lingelbach S, Jaramillo JC. Safety and immunogenicity of a live-attenuated chikungunya virus vaccine in adolescents: final results from a 12-month, double-blind, randomised, placebo-controlled, phase 3 trial in endemic areas of Brazil. Lancet Infect Dis. 2025 Dec 8:S1473-3099(25)00631-0. doi: 10.1016/S1473-3099(25)00631-0. Online ahead of print. PMID 41380703
- [Derived] Buerger V, Hadl S, Schneider M, Schaden M, Hochreiter R, Bitzer A, Kosulin K, Mader R, Zoihsl O, Pfeiffer A, Loch AP, Morandi E Jr, Nogueira ML, de Brito CAA, Croda J, Teixeira MM, Coelho IC, Gurgel R, da Fonseca AJ, de Lacerda MVG, Moreira ED Jr, Veiga APR, Dubischar K, Wressnigg N, Eder-Lingelbach S, Jaramillo JC. Safety and immunogenicity of a live-attenuated chikungunya virus vaccine in endemic areas of Brazil: interim results of a double-blind, randomised, placebo-controlled phase 3 trial in adolescents. Lancet Infect Dis. 2025 Jan;25(1):114-125. doi: 10.1016/S1473-3099(24)00458-4. Epub 2024 Sep 5. PMID 39243794